CLINICAL TRIAL: NCT00605852
Title: A Double-blind, Placebo-controlled, Randomized Cross-over Single Dose Escalation Study and a Double-blind, Placebo-controlled, Randomised Parallel Group 7-days Once Daily Repeat Dose Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral H1/H3 Dual Antagonist Compound in Healthy Male Subjects
Brief Title: Investigation Of a New Oral Anti-Histamine in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: HH3110161
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Allergic rhinitis; first time in human
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — GSK 835726

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Subjects receiving treatment in cohort I (Experimental): Eligible subjects will receive three single doses of GSK835726 and one single dose of placebo in cohort I.
  Interventions: Drug: GSK835726; Drug: Placebo
- Subjects receiving GSK835726 in cohort II (Experimental): Eligible subjects will receive repeat doses of GSK835726 once daily for 7 days.
  Interventions: Drug: GSK835726
- Subjects receiving placebo in cohort II (Placebo Comparator): Eligible subjects will receive repeat doses of placebo once daily for 7 days.
  Interventions: Drug: Placebo
- Subjects receiving treatment in cohort III (Experimental): Eligible subjects will receive two single doses of GSK835726 and one single dose of placebo in cohort III.
  Interventions: Drug: GSK835726; Drug: Placebo

INTERVENTIONS:
Drug: GSK835726 — GSK835726 will be available in single dose and repeat dose formulations.
  Arms: Subjects receiving GSK835726 in cohort II; Subjects receiving treatment in cohort I; Subjects receiving treatment in cohort III
Drug: Placebo — Placebo will be given to subjects.
  Arms: Subjects receiving placebo in cohort II; Subjects receiving treatment in cohort I; Subjects receiving treatment in cohort III

SUMMARY:
This study is designed to assess the safety and tolerability of single, escalating oral doses and repeat oral doses (7 days, once daily) of GSK835726 in healthy male subjects

DETAILED DESCRIPTION:
A double-blind, placebo controlled, randomized cross-over single dose escalation study and a double-blind, placebo controlled, randomised parallel group 7-days once daily repeat dose study to investigate safety, tolerability, pharmacokinetics and pharmacodynamics of oral H1/H3 dual antagonist compound in healthy male subjects

ELIGIBILITY:
Inclusion criteria:

* Male aged between 18 and 50 years inclusive.
* Body mass index within the range 19-29kg/m2 (inclusive), with weight range of 55kg-100kg (inclusive).
* Healthy (defined as individuals who are free from significant nasal, cardiac, pulmonary, gastrointestinal, hepatic, renal, haematological, malignancy, endocrine, neurological and psychiatric disease as determined by history, physical examination and screening investigations).
* Non-smoking status as verified by urinary cotinine levels below 300 ng/mL cotinine at the screening visit. This can include ex-smokers who have given up smoking for >1 year.
* Subjects to be entered in cohorts I and III only: Skin prick test reactivity to histamine of 3mm wheal > than saline control and some associated surrounding erythema.
* Subjects to be entered in cohorts I and III only: Negative skin prick test reactivity to saline control.
* The subject is able and willing to give written informed consent to take part in the study and is available to complete all study measurements.
* If sexually active, male subjects must agree to use a condom with spermicide during sexual intercourse, from the first dose of the study drug until 84 days after the last dose. In addition, female partners of male subjects, who are of childbearing potential, must use a reliable contraceptive method or they must refrain from sexual intercourse from the first dose of study medication until 84 days after the last dose. Reliable forms of contraception include an IUD, condom or diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants, contraceptive patches or a tubal ligation."

Exclusion criteria:

* As a result of the medical interview, physical examination or screening investigations, the Investigator or appropriately qualified designee considers the subject unfit for the study.
* The subject has a history of drug or any other allergy, which, in the opinion of the Investigator or appropriately qualified designee, contraindicates their participation, including known or suspected personal history or family history of adverse reactions or hypersensitivity to anti histamines.
* The subject has participated in a study with a new molecular entity during the previous 3 months or any other study during the previous 2 months.
* The subject regularly, or on average, drinks more than 21 units of alcohol a week or more than an average intake of 3 units per day (One unit = 125ml wine or 25ml spirits or 250ml normal strength lager).
* The subject is currently taking regular (or a course of) medication, prescribed (including all anti-allergy medication) or not (including over the counter medication or herbal remedies such as St Johns Wort). Paracetamol is an exception and will be permitted at daily doses of up to 4g following all doses of investigational product.
* The subject has tested positive for hepatitis C antibody or hepatitis B surface antigen.
* The subject has tested positive for HIV.
* The subject has a positive drugs of abuse and alcohol test.
* Donation of blood (450 mL or more) within 2 months of screening.
* Donation during the study would result in >500mL of blood being donated over a 56 day period
* Significant cardiac conduction abnormalities on two or more ECG tracings separated by at least 5 minutes at screening, including:

  * QTc interval > 450 msec
  * PR interval > 240 msec
  * Evidence of second- or third- degree atrioventricular (AV) block
  * Ventricular rate < 45 beats per minute (bpm) or > 100 bpm
  * Pathological Q-waves (defined as Q-wave > 40 msec or depth greater than 0.4-0.5 mV)
  * Evidence of ventricular pre-excitation
  * Evidence of left axis deviation, non-specific intraventricular conduction delay (QRS duration > 120 msec), or complete left bundle branch block
* Subjects with Perennial Allergic Rhinitis (PAR) and Seasonal Allergic Rhinitis (SAR), unless subjects with SAR are asymptomatic and it is outside of the pollen season
* Subjects with dermatographism and other skin conditions that might interfere with the wheal and flare test.
* Subjects who are unable to comply with study procedures.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2007-10-29 (Actual); Primary Completion 2008-05-03 (Actual); Study Completion 2008-05-03 (Actual)

PRIMARY OUTCOMES:
ECG monitoring during 24 hours after each dose in the single dose cohorts and on days 1 and 7 in the repeat dose cohorts. | during 24 hours after each dose in the single dose cohorts and on days 1 and 7 in the repeat dose cohorts.
Heart rate and blood pressure changes over 24 hours after dosing in single and repeat dose cohorts | over 24 hours after dosing in single and repeat dose cohorts

SECONDARY OUTCOMES:
Change in plasma drug concentration (AUC, Cmax, t1/2, tmax) | over 24 hours after dosing
Changes in histamine-induced wheal and flare measurements | over 24 hours after dosing
Derived pharmacokinetic parameters for GSK835726 including area under the plasma drug concentration versus time curve (AUC(0-t), AUC(0-¥)), maximum observed plasma drug concentration (Cmax), | over 24 hours after dosing
time to maximum observed plasma drug concentration (tmax), apparent clearance (CL/F) and terminal half life (t1/2) following single and repeat oral dosing. | over 24 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Daley-Yates P, Ambery C, Sweeney L, Watson J, Oliver A, McQuade B. The efficacy and tolerability of two novel H(1)/H(3) receptor antagonists in seasonal allergic rhinitis. Int Arch Allergy Immunol. 2012;158(1):84-98. doi: 10.1159/000329738. Epub 2011 Dec 29. PMID 22212854
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study HH3110161 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/HH3110161?search=study&study_ids=HH3110161#rs
- Available data/document: Annotated Case Report Form: HH3110161 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: HH3110161 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: HH3110161 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: HH3110161 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: HH3110161 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: HH3110161 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: HH3110161 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register